CLINICAL TRIAL: NCT06934629
Title: Effect of Tecar Therapy During Active Exercises on Dynamic Balance in Acute Ankle Sprain
Brief Title: Efficacy of Tecar Device With Exercises in Ankle Sprain
Acronym: TECAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Morsy Elsayed Ali Morsy, resident physiotherapist registered for master degree, Cairo University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005596
Record Dates: First submitted 2025-04-02; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Ankle Sprain; TECAR Therapy; TECAR Therapy Efficacy in the Treatment of Ankle Sprain; Ankle Dynamic Balance; Ankle Pain; Ankle Proprioception
Keywords: Ankle pain; ankle dynamic balance; Ankle proprioception; Ankle daily function; TECARtherapy
MeSH Terms: conditions — Ankle Injuries | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Treatment will be for 4 weeks with 2 sessions per week. TECAR application will be 20 mins per session (10 mins capacitive and 10 mins resistive) during ankle and subtalar ROM in a pain-free range, calf muscle stretch, ankle strengthening exercises against resistance bands in all directions, weight-bearing exercise, forward lunges, bilateral and unilateral squats, bilateral and unilateral heel raises against bodyweight resistance, and balance training.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TECAR therapy group (Experimental): traditional therapeutic exercises for ankle sprain and TECAR therapy application during exercises .
  Interventions: Device: TECAR therapy
- Conventional therapy group (Active Comparator): traditional therapeutic exercises for ankle sprain
  Interventions: Other: therapeutic exercises

INTERVENTIONS:
Device: TECAR therapy — TECAR application will be 20 mins per session (10 mins capacitive and 10 mins resistive) during ankle and subtalar ROM in a pain-free range, calf muscle stretch, ankle strengthening exercises against resistance bands in all directions, weight-bearing exercise, forward lunges, bilateral and unilateral squats, bilateral and unilateral heel raises against bodyweight resistance, and balance training.
  Arms: TECAR therapy group
Other: therapeutic exercises — the conventional therapy which is ankle and subtalar ROM in a pain-free range, calf muscle stretch, ankle strengthening exercises against resistance bands in all directions, weight-bearing exercise, forward lunges, bilateral and unilateral squats, bilateral and unilateral heel raises against bodyweight resistance, and balance training.
  Arms: Conventional therapy group

SUMMARY:
The goal of this clinical trial is to evaluate the effect of applying TECAR therapy during active therapeutic exercises on pain, ankle dynamic balance, proprioception, and daily function in patients with acute ankle sprain.

the main questions it aims to answer are:

* Does there is a significant effect of applying TECAR therapy during active exercise after acute lateral ankle sprain on Pain?
* Does there is a significant effect of applying TECAR therapy during active exercise after acute lateral ankle sprain on balance?
* Does there is a significant effect of applying TECAR therapy during active exercise after acute lateral ankle sprain on proprioception?
* Does there is a significant effect of applying TECAR therapy during active exercise after acute lateral ankle sprain on daily function? The patients will be randomly divided into two groups. The control group (A) will receive the conventional therapy which is ankle and subtalar ROM in a pain-free range, calf muscle stretch, ankle strengthening exercises against resistance bands in all directions, weight-bearing exercise, forward lunges, bilateral and unilateral squats, bilateral and unilateral heel raises against bodyweight resistance, and balance training. The experiment group (B) will receive conventional therapy with TECAR therapy application during active therapeutic exercises.

Treatment will be for 4 weeks with 2 sessions per week. TECAR application will be 20 mins per session (10 mins capacitive and 10 mins resistive).

To the best of the researchers' knowledge, no study has proved the effects of applying TECAR therapy during active therapeutic exercises after an acute lateral ankle sprain has yet been done. Thus, the purpose of the present study was to prove if there an effect of applying TECAR therapy during active therapeutic exercises included in the conventional physiotherapy (PRICE with therapeutic exercises) and conventional physiotherapy alone on pain, ankle dynamic balance, proprioception, and daily function in subjects with an acute lateral ankle sprain.

ELIGIBILITY:
Inclusion Criteria:

* Gender will be male and female.
* Age from 20-40 years old.
* Grade | and || lateral ankle sprain.
* Patients who will be diagnosed and referred by orthopedic surgeon.
* acute stage of lateral ankle sprain.
* BMI ≤ 30.
* Positive confirming tests.

Exclusion Criteria:

* Ankle fractures such as talus bone fracture, tibia fracture, ankle dislocation.
* Unwilling to continue treatment.
* Contraindications to use TECAR therapy, such as pregnancy, the presence of malignant tissue, tumors, in the ankle, and electrical devices implanted in the body.
* Grade ||| ankle sprain.
* Systematic diseases such as rheumatoid arthritis.
* Recently received intra-steroid injection
* Pain exacerbation during the intervention.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
1.ankle dynamic balance. | from enrollment to the end of treatment at 4 weeks.
  using Star Excursion Balance Test
2.pain | from enrollment to the end of treatment at 4 weeks.
  using Numerical pain rating scale (NPRS)

SECONDARY OUTCOMES:
3. proprioception | from enrollment to the end of treatment at 4 weeks.
  using digital inclinometer

CONTACTS AND LOCATIONS:
Locations (1):
- Andalusia hospital in Alexandria, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided